CLINICAL TRIAL: NCT02566122
Title: Establishment of Normal Muscle Strength Measured by Hand-held Dynamometer and Muscle Mass Assessed by Ultrasonography for French Population
Brief Title: Establishment of Normal Muscle Strength for French Population
Status: Terminated | Type: Observational
Why Stopped: not enough patients
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5423
Record Dates: First submitted 2013-02-12; First posted 2015-10-02 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Muscle Mass; Muscle Strength
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- muscle strength ,muscle mass
  Interventions: Other: measurements

INTERVENTIONS:
Other: measurements

SUMMARY:
Normal values for muscle strength using hand held dynamometer and muscle mass using echography are largely unknown. The objective of the present study is to establish normal values of these measurements in population living in France.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-90 years

Exclusion Criteria:

* Patients < 20 years and > 90 years,
* Athletes involved in international sport competition
* Rheumatic or neuromuscular disease
* Other decompensated pathological conditions
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: male and female volunteers aged 18-90 years
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
measuring muscle mass using echography | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'exploration fonctionnelle Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace, France